CLINICAL TRIAL: NCT05721339
Title: Impact of Virtual Group-Based Acceptance and Commitment Therapy on Social Adjustment and Work-Family Conflict Among Intern Nurses: A Randomized Control Trial
Brief Title: Virtual Acceptance and Commitment Therapy Impact on Social Adjustment and Work-Family Conflict Among Intern Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, ayman el-ashry, lecturer at psychiatric and mental health nursing, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00013620-50-9-2022
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Nurse's Role
Keywords: Acceptance and Commitment Therapy; Intern Nurses; Social Adjustment; Work-Family Conflict
MeSH Terms: conditions — Social Adjustment | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and commitment therapy (Experimental): Intern nurses will participate in acceptance and commitment therapy through virtual group-based eight sessions twice weekly with homework assignments between sessions and skills demonstration.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- control group (No Intervention): Intern nurses who will not participate in acceptance and commitment therapy. And they are undergoing the pre-and post-tests and the post-test follow-up test.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — ACT will be applied through 8 sessions by the psychological flexibility processes, which were grouped into three response styles: open, aware, and active. Openness is reflected by acceptance, which means the conscious embrace of psychological events without unnecessary attempts to change their frequency. Defusion means untangling unhelpful thoughts and responding to mental experiences as experiences rather than guides to action. The awareness set, which is reflected by applying self-as-context, which means a continuous and secure "I" from which events are experienced but distinct from those events. A present moment means ongoing, nonjudgmental contact with internal and external events as they occur in the present moment. The active set, which was reflected by making the intern nurses embrace their desired and chosen life values directions, and commit action to selected values.
  Other Names: functional contextualism
  Arms: Acceptance and commitment therapy

SUMMARY:
Work and family are the two most influential aspects of a person's life. The conflict between work and family can adversely affect an organization's and an individual's health and well-being. Research is necessary to describe, understand, and address work-family conflict because it arises from how people perceive it. Studies on social adjustment for healthcare staff and nursing interns are scarce in Egypt, according to researchers. Recently, ACT has been utilized to treat various psychological issues and challenges at work, among others. Therefore, the present study aimed to evaluate the impact of virtual group-based acceptance and commitment therapy on intern nurses' social adjustment and work-family conflict.

Research Hypothesizes Intern nurses who engaged in a virtual group-based acceptance and commitment therapy will exhibit lower level of family-work conflict than the control group.

Intern nurses who engaged in a virtual group-based acceptance and commitment therapy will exhibit a higher level of social adjustment than the control group.

DETAILED DESCRIPTION:
Given the nature of the nursing profession, intern-nurses frequently interact with patients, their families, physicians, and all levels of hospital administration. Time, long-term work, shifting hours, sleeplessness, death observation, cancer, high healthcare demands, and a low tolerance for incompetence are all sources of stress for those newly graduate nurses. As a result, their social adjustment significantly affects whether they are able to remain motivated and collaborative. Work conflict has become a type of intra-role conflict in which both parties' work and family responsibilities overlap. This term applies to the unfavorable interaction that exists between work and family when there is a discrepancy between reality and expectations, which disrupts and affects job performance at work or at home.

Intern nurses was trained in the Main University Hospital (El-Miri), University Hospital Smouha, El Shatby Hospital for Obstetricians and Gynecologists, and El Hadara Orthopedic and Traumatology University hospital this study will be conducted. These hospitals were affiliated to Alexandria University for clinical training of intern-nurses in all nursing disciplines for around 12 months, beginning in September 2022 and ending in August 2023.According to the records of the internship candidates' affairs department and internship coordinator at the Faculty of Nursing, the total number of enrolled candidates during this academic year was 800 candidates. G*Power Windows 3.1.9.7 a program with the following parameters was used to estimate the participants: Power (1-β err prob) =.88, effect size =.5, α err prob = .05. The program identified a minimum sample size of 34 intern nurses for each group. Thus, the sample will be comprised of 70 intern nurses, the study group will compose of n = 35 participants, the control group will be the same number. A representative sample of intern nurses will be allocated to either the study or control groups using the random assignment technique.

"Implementation phase": Seventy intern-nurses will be selected at random to assign the study or control group, the researchers will attempt to match the control group as accurately as possible in terms of age, gender, marital status, and working hours' duration. Then, those participants will meet individually in a private online meeting to create rapport, discuss the goal of the study and the therapy that will be employed, and obtain their written consent.

The pretest phase will begin with the collection of baseline assessment data from the study and control groups on the study instruments II, III, and IV, utilizing computerized forms.

The intervention phase will start with the study group being randomly will be divided into five small groups, each having six ACT participants.

For three weeks, the ACT sessions will be held twice a week for 90 minutes each. Each session will be conducted by two researchers, one as a leader to explain the fundamental core of the therapy for about 60 minutes and the other as a mediator to organize homework assignments with the participants and answer any queries for about 30 minutes.

Evaluation or Follow-up Phase." The last phase, "the posttest," will be done twice immediately following the end of all sessions, as well as a one-month later as a follow-up utilizing tools II, III and V.

ELIGIBILITY:
Inclusion Criteria:

* The beginner intern nurses at the academic year 2022-2023.
* Single candidates.
* Willing to participate in the study.

Exclusion Criteria:

* Intern nurses who diagnosed with any chronic medical diseases.
* Intern nurses who diagnosed with any mental illnesses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
The Work-related Acceptance and Action Questionnaire | up to 14 weeks
  It was developed to assess psychological flexibility in professional contexts. It consists of seven statements assessed on a Likert Scale from 1 (Never true) to 7 (Always true), such as "I can admit my faults at work and yet be successful," and "I can work efficiently even when I doubt myself." The items stand for people's ability to take goal-directed action in the face of unpleasant internal experiences. The Work-related Acceptance and Action Questionnaire scores range from 7 to 49, with higher scores suggesting greater psychological flexibility.
The Social Adjustment Scale-Self Report | up to 14 weeks
  The Social Adjustment Scale-Self Report is a popular 54-items self-reported social adjustment scale that assesses instrumental and expressive role performance over the previous two weeks. It addresses six areas of functioning: employment (as a paid worker, unpaid homemaker, or student), social and leisure activities, interactions with extended family, marital partner role, parenting role, and role within the family unit.The elements in each of the six categories encompass four sorts of content: performance at anticipated tasks, interpersonal friction, finer characteristics of interpersonal relationships, and emotions and satisfactions. The full-length Social Adjustment Scale-Self Report takes around 15-20 minutes to administer.The higher the score of Social Adjustment Scale-Self Report, the more impairment in social adjustment.
Work-Family Conflict Scale | up to 14 weeks
  Work-family conflict and family-work conflict were divided on the scale. Each subscale comprised five items that measured the level of conflict in that subscale. It is evaluated on a 7-point Likert scale, with 1 being "very strongly disagree" and 7 being "very strongly agree". The items for each subscale are totaled to supply the overall scores of Work-Family Conflict Scale (ranging from 7 to 35) and Family-Work Conflict Scale (ranging from 7 to 35); higher scores show higher degrees of conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M El-Ashry, PHD, Principal Investigator — Faculty of nursing, Alexandria University, Egypt
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prudenzi A, Graham CD, Flaxman PE, Wilding S, Day F, O'Connor DB. A workplace Acceptance and Commitment Therapy (ACT) intervention for improving healthcare staff psychological distress: A randomised controlled trial. PLoS One. 2022 Apr 20;17(4):e0266357. doi: 10.1371/journal.pone.0266357. eCollection 2022. PMID 35442963
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] AlAzzam M, AbuAlRub RF, Nazzal AH. The Relationship Between Work-Family Conflict and Job Satisfaction Among Hospital Nurses. Nurs Forum. 2017 Oct;52(4):278-288. doi: 10.1111/nuf.12199. Epub 2017 Apr 13. PMID 28407250
- [Derived] El-Ashry AM, Elhay ESA, Taha SM, Salem ESAEHES, El-Sayed MM. Impact of virtual group-based acceptance and commitment therapy on social adjustment and work-family conflict among intern nurses: a randomized control trial. BMC Psychiatry. 2023 Aug 1;23(1):552. doi: 10.1186/s12888-023-05045-8. PMID 37525125
- See also: a worldwide online learning and research community, and a living resource for anyone interested in Acceptance and commitment therapy and Contextual Behavioral Science. — https://contextualscience.org/